CLINICAL TRIAL: NCT01613469
Title: Maintenance of Chemotherapy Following Neoadjuvant Chemoradiation Therapy for Distal Rectal Cancer
Brief Title: Maintenance Chemotherapy After Neoadjuvant Chemoradiation Therapy for Distal Rectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Re-eval of patient population
Sponsor: Marks, John, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R12-3092L
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Rectal Neoplasms
Keywords: fluorouracil; leucovorin; radiotherapy; neoadjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5FU/Leucovorin- post distal rectal srgy (Other): Assess complete clinical response rate following neoadjuvant chemoradiation in patients with distal rectal cancer
  Interventions: Drug: 5FU/Leucovorin

INTERVENTIONS:
Drug: 5FU/Leucovorin — 450 mg/m2 of 5-FU plus 50 mg Leucovorin given in 3 cycles during radiation (one cycle is the administration every day for 3 consecutive days, a cycle is 21 days)followed by 450 mg/m2 of 5-FU plus 50 mg Leucovorin given in 3 cycles after completion of radiation.
  Other Names: SOC intervention

SUMMARY:
This study will assess the complete clinical response (no clinical evidence of remaining disease or recurrence of disease)in rectal cancer that arises within 3 inches of the anal opening after radiation therapy given at the same time as chemotherapy over a 6 week period, followed by chemotherapy alone given three times over an additional 9 weeks. Follow-up begins with an examination at the end of treatment (at 15 weeks), with ongoing follow-up every 4-6 weeks for one year.

DETAILED DESCRIPTION:
Research has shown that low rectal cancer treated with neoadjuvant chemoradiation (54Gy concurrent with 3 cycles of 5-FU/Leucovorin) followed by 3 additional cycles of 5FU/Leucovorin, followed by close follow-up (every 4-6 weeks for one year)has had good success in achieving complete clinical response, avoiding surgical intervention. If at follow-up remaining disease is found or if there is recurrent disease, surgery can be performed.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* tumor potentially resectable en bloc; tumors tethered or fixed to a structure that can be removed
* clinical/radiological stages T2,T3,or T4, N0-1
* ANC >1500, PLT>100,000
* AST and alkaline phosphatase < 2.5 X ULN
* bilirubin < 1.5 X ULN
* CrCl > 50 ml/min using Cockcroft-Gault formula
* KPS >60
* ECOG Performance Scale 0-2
* No malignancies within previous 5 years other than non-melanoma skin cancer, in-situ cervical cancer, in-situ ductal breast cancer
* no evidence of metastatic disease

Exclusion Criteria:

* initial tumor fixation to pelvic bone or side wide; technically unresectable disease
* any evidence of distant metastasis
* perforation
* obstruction
* hereditary non-polyposis colorectal cancer
* synchronous primary colon carcinomas except T1 lesions
* known dihydropyrimidine dehydrogenase deficiency
* prior radiation therapy to the pelvis
* prior chemotherapy for malignancies
* known existing uncontrolled coagulopathy
* pregnancy or lactation
* women of childbearing potential not using reliable and appropriate contraceptive method
* serious, uncontrolled concurrent infection(s)
* participation in any investigational drug study within 4 weeks preceding the start of study treatment
* clinically significant heart disease
* other serious uncontrolled medical conditions that might compromise study participation (in the investigator's opinion)
* major surgery within 4 weeks prior to the study treatment
* lack of physical integrity of the upper GI tract or malabsorption syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-08; Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
To assess the complete clinical response rate following neoadjuvant chemoradiation in patients with distal rectal cancer. | One year from the time of chemoradiation
  Primary endpoints are the proportion of subjects with complete clinical response to chemoradiation therapy at no sooner than 9 weeks from treatment completion, and maintenance of continuous freedom from local failure for one year.

SECONDARY OUTCOMES:
The proportion of subjects with complete pathological response at surgical resection | One year from chemoradiation therapy
  At surgical intervention for incomplete clinical response or recurrence, complete pathological response is no evidence of residual disease at pathological examination of the resected specimen.

CONTACTS AND LOCATIONS:
Overall Officials: John Marks, MD, Principal Investigator — Main Line Health
Locations (1):
- Lankenau Medical Center, Wynnewood, Pennsylvania, United States

REFERENCES:
- [Background] Habr-Gama A, Perez RO, Kiss DR, Rawet V, Scanavini A, Santinho PM, Nadalin W. Preoperative chemoradiation therapy for low rectal cancer. Impact on downstaging and sphincter-saving operations. Hepatogastroenterology. 2004 Nov-Dec;51(60):1703-7. PMID 15532809
- [Background] Habr-Gama A, de Souza PM, Ribeiro U Jr, Nadalin W, Gansl R, Sousa AH Jr, Campos FG, Gama-Rodrigues J. Low rectal cancer: impact of radiation and chemotherapy on surgical treatment. Dis Colon Rectum. 1998 Sep;41(9):1087-96. doi: 10.1007/BF02239429. PMID 9749491
- [Background] Habr-Gama A, Perez RO, Nadalin W, Nahas SC, Ribeiro U Jr, Silva E Sousa AH Jr, Campos FG, Kiss DR, Gama-Rodrigues J. Long-term results of preoperative chemoradiation for distal rectal cancer correlation between final stage and survival. J Gastrointest Surg. 2005 Jan;9(1):90-9; discussion 99-101. doi: 10.1016/j.gassur.2004.10.010. PMID 15623449
- [Background] Habr-Gama A, Perez RO, Sabbaga J, Nadalin W, Sao Juliao GP, Gama-Rodrigues J. Increasing the rates of complete response to neoadjuvant chemoradiotherapy for distal rectal cancer: results of a prospective study using additional chemotherapy during the resting period. Dis Colon Rectum. 2009 Dec;52(12):1927-34. doi: 10.1007/DCR.0b013e3181ba14ed. PMID 19934911
- [Background] Habr-Gama A, Perez RO. Non-operative management of rectal cancer after neoadjuvant chemoradiation. Br J Surg. 2009 Feb;96(2):125-7. doi: 10.1002/bjs.6470. No abstract available. PMID 19160360
- [Background] Petersen S, Hellmich G, von Mildenstein K, Porse G, Ludwig K. Is surgery-only the adequate treatment approach for T2N0 rectal cancer? J Surg Oncol. 2006 Apr 1;93(5):350-4. doi: 10.1002/jso.20452. PMID 16550556